CLINICAL TRIAL: NCT01587846
Title: Lactobacillus Reuteri in Treatment of Functional Abdominal Pain and Chronic Constipation in Children - Randomized, Double Blind, Placebo Controlled Study
Brief Title: Lactobacillus Reuteri in Treatment of Functional Abdominal Pain and Chronic Constipation in Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sisters of Mercy University Hospital (Other)
Collaborators: BioGaia AB (Industry)
Responsible Party: Principal Investigator, Sanja Kolacek, MD, PhD, Head of the Department of Pediatrics, Clinical Professor, Principal Investigator, Sisters of Mercy University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LR-2012-KL
Record Dates: First submitted 2012-04-23; First posted 2012-04-30 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Abdominal Pain; Constipation - Functional
Keywords: abdominal pain, constipation, Lactobacillus reuteri
MeSH Terms: conditions — Abdominal Pain; Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Probiotic/abdominal pain (Experimental): Children with functional abdominal pain that will receive probiotic.
  Interventions: Dietary Supplement: Administration of L.reuteri in children with abdominal pain
- Placebo/abdominal pain (Experimental): Children with functional abdominal pain that will receive placebo.
  Interventions: Dietary Supplement: Administration of placebo in children with abdominal pain
- Probiotic/constipation (Experimental): Children with chronic constipation tha will receive probiotic plus lactulose
  Interventions: Dietary Supplement: Administration of L.reuteri in children with constipation
- Placebo/chronic constipation (Experimental): Children with chronic constipation that will receive placebo plus lactulose
  Interventions: Dietary Supplement: Administration of placebo in children with constipation

INTERVENTIONS:
Dietary Supplement: Administration of L.reuteri in children with abdominal pain — Group of around 75 children which will receive L. reuteri at a dose 100.000.000 CFU per dose for 3 months. The active study product consists of a citrus flavored 450 mg chewable tablet containing freeze-dried L. reuteri DSM 17938. The study product is a convex tablet 10.3 mm in diameter, plain on both sides and with faint spots. It is composed of freeze-dried L. reuteri, isomalt, xylitol, sucrose distearate, hydrogenated palm oil, lemon-lime flavoring and anhydrous citric acid. The total viable count of L. reuteri is 1x100.000.000 live bacteria (CFU)/tablet.
  Arms: Probiotic/abdominal pain
Dietary Supplement: Administration of placebo in children with abdominal pain — Group of around 75 children which will receive placebo for 3 months. The placebo consists of a citrus flavored 450 mg chewable convex tablet 10.3 mm in diameter, plain on both sides and with faint spots. It is composed of isomalt, xylitol, sucrose distearate, hydrogenated palm oil, lemon-lime flavoring and anhydrous citric acid.
  Arms: Placebo/abdominal pain
Dietary Supplement: Administration of L.reuteri in children with constipation — Group of around 75 children which will receive L. reuteri at a dose 100.000.000 CFU per dose plus lactulose in a dose 1-3 ml/kg, according to the stool frequency and consistency, for 3 months. The active study product consists of a citrus flavored 450 mg chewable tablet containing freeze-dried L. reuteri DSM 17938. The study product is a convex tablet 10.3 mm in diameter, plain on both sides and with faint spots. It is composed of freeze-dried L. reuteri, isomalt, xylitol, sucrose distearate, hydrogenated palm oil, lemon-lime flavoring and anhydrous citric acid. The total viable count of L. reuteri is 1x100.000.000 live bacteria (CFU)/tablet.
  Arms: Probiotic/constipation
Dietary Supplement: Administration of placebo in children with constipation — Group of around 75 children which will receive placebo plus lactulose in a dose 1-3 ml/kg, according to the stool frequency and consistency, for 3 months. The placebo study product consists of a citrus flavored 450 mg chewable convex tablet 10.3 mm in diameter, plain on both sides and with faint spots. It is composed of isomalt, xylitol, sucrose distearate, hydrogenated palm oil, lemon-lime flavoring and anhydrous citric acid.
  Arms: Placebo/chronic constipation

SUMMARY:
Beneficial therapeutic effect of probiotics has been reported in children with irritable bowel syndrome, but not consistently in other functional gastrointestinal disorders. Although there is evidence that probiotics increase stool frequency and decrease stool consistency in healthy individuals the evidence for efficacy in constipation is limited.

Children with functional abdominal pain (FAP) and constipation will be included in the study. Children with FAP will be randomized in one of two groups and will receive either L. reuteri in a daily dose of 108 CFU, or placebo during three months. Children with chronic constipation will receive either L. reuteri in a daily dose of 108 CFU and lactulose, or placebo and lactulose. Frequency and intensity of episodes of abdominal pain during and after intervention will be recorded in children with FAP. Frequency of defecation, stool consistency and need for lactulose will be recorded in children with chronic constipation.

DETAILED DESCRIPTION:
Part I. Lactobacillus reuteri in treatment of functional abdominal pain in children

1. Introduction

   Probiotics are defined as live microorganisms which confer a beneficial health effect on a human host. Their beneficial effects are based on: promotion of resistance to enteric pathogens, prevention of small bowel bacterial overgrowth and immune system modulation. The most commonly used probiotics are bacteria of genera Lactobacillus or Bifidobacterium. Other nonpathogenic genera, including Escherichia, Enterococcus and Bacillus, and nonbacterial organisms, such as a nonpathogenic yeast Saccharomyces boulardii, have also been studied.

   A probiotic preparation must contain a certain minimum number of colony-forming units (CFU) per dose (4). Doses used in therapeutic and preventive trials vary. A daily intake of 1.000.000 to 1.000.000.000 CFUs is a reported minimum for therapeutic purposes. There is an increasing number of studies on beneficial effects of probiotics in treatment of acute infectious diarrhoea, and prevention of antibiotic associated diarrhoea. Role of probiotics in the treatment of functional GI disorders is still controversial.

   Recurrent or chronic abdominal pain affects 10-15% of school-age children. Functional abdominal pain (FAP) is defined as occasional or continuous abdominal pain with a frequency of at least once a weak during at least two months; most frequently the pain is located around umbilicus and not related to meals. Although visceral hypersensitivity plays a certain role in pathogenesis of a pain, FAP is probably a complex disorder. Irritable bowel syndrome is defined as abdominal pain or discomfort associated (in at least 25% of time) with two of these criteria: 1) relief after defecation, 2) change in stool frequency or 3) change in stool consistence.

   Pathogenesis of this disorder is complex and included interaction of psychosocial factors, motility disorder and visceral hypersensitivity. Therapeutic possibilities are pepermint oil, serotonin reuptake inhibitors and tricyclic antidepressants. Although there are studies confirming positive effect of probiotics in children and adults with IBS, there is no clear evidence for the effect of probiotics in FAP. The number of studies and the patients included is also relatively small to draw final conclusions.

   Therefore, the aim of this study is to investigate whether Lactobacillus reuteri could have a beneficial role in treatment of functional abdominal pain in children.
2. Study population

   All paediatric patients referred to a pediatric gastroenterologist for functional abdominal pain (age 4-18 years) at the Department of Paediatrics, Children's Hospital Zagreb, University Hospital "Sestre Milosrdnice".

   Their symptoms will be evaluated with the use of Rome III criteria for functional gastrointestinal disorders of children and visual-analogue scale (Wong-Baker faces pain rating scale) for pain.
3. Intervention

   All children with functional abdominal pain whose parents have signed an inform consent; will receive either probiotic or placebo for 3 months.

   As a part of randomized, double blind controlled trail, patients will be randomized into one group (A or B) and none of investigators or patients will know true nature of the product (active product or placebo).
4. Hypothesis

   L. reuteri can effectively treat functional abdominal pain in children.
5. Aims

   To evaluate the effect of L. reuteri on the number and severity of episodes pain in children with functional abdominal pain
6. Sample size for independent cohort study

   Probability of event in control group = 0,5 Difference between groups: 30% (ref. 18) Probability of event in experimental group = 0,35 Controls per case subject = 1 Alpha = 0,05 Power = 0,95

   For Fisher's exact tests:

   N (total) = 2x138 (69 per group)
7. Randomization

The trial will be prospective, randomized, double blind, placebo controlled study. Probiotics, Lactobacillus reuteri and placebo will be supplied by Biogaia, Stockholm, Sweden.

Randomization will be performed using computer generated numbers based on which every patient will get a number and receive the preparation successively. All products, probiotic and placebo will be packed in identical packages and will have identical smell and taste and have only mark "A" or "B", true nature of the preparation would not be revealed to investigators or to participants.

After all calculations and statistical analysis true nature of the preparations will be revealed in front of uninvolved witnesses.

BASELINE (VISIT 1): randomization VISIT 2: 4 weeks after randomization END OF STUDY (VISIT 3): End of study 3 months after baseline VISIT 4: 4 weeks after the end of study (16 weeks after the baseline).

All the symptoms will be monitored using diaries attached to protocol.

In order to achieve adherence to therapeutic protocol parents will be contacted by phone at least once in 7-10 days. Participants will be instructed to keep diary on a daily basis (adherence to therapy, pain diary). All patients will return packages with all used, and unused product.

Part II. Lactobacillus reuteri in treatment of chronic constipation in children - randomized, double blind, placebo controlled study

1. Introduction

   Defecation disorder is a frequent problem in childhood and in 90-95% of children presents a functional problem.

   Chronic constipation in childhood is defined with at least two of these criteria: 1) stools twice a weak of rarer, 2) at least one episode of fecal incontinence per weak after having already achieved toilet control, 3) stool withholding manoeuvres, 4) painful of difficult defecation, 5) presence of large fecal masses in rectum, 6) stool of a large caliber.

   In adults, there is some evidence that chronic constipation is related to a gastrointestinal flora with decreased number of lactobacilli and bifidobacteria and increased potentially pathogenic bacteria, yeast and fungi. Dysbiosis with increased clostridia has also been reported in children with chronic constipation. Majority of infants have higher frequency of defecation and the consistency of stools is softer in breast-fed infants in first months of life. Breast-fed babies produce more lactic acid in colon which decreases intestinal pH. As a result bifidobacteria proliferate. Also, colonic flora has been shown to influence peristalsis. Although there is evidence that lactobacilli and bifidobacteria increase stool frequency and decrease stool consistency in normal individuals the evidence for efficacy in constipation is limited.

   Therefore, the aim of this study is to investigate whether Lactobacillus reuteri could have a beneficial role in treatment of chronic constipation in children.
2. Study population

   All paediatric patients referred to a pediatric gastroenterologist for chronic constipation (age 2-18 years) at the Department of Paediatrics, Children's Hospital Zagreb, University Hospital "Sestre Milosrdnice".

   Their symptoms will be evaluated with the use of Rome III criteria for functional gastrointestinal disorders of children, Bristol scale for stool shape and consistence and visual-analogue scale (Wong-Baker faces pain rating scale) for pain.
3. Intervention

   All children with chronic constipation whose parents have signed an inform consent; will be randomly assigned into one of two following groups: probiotic or placebo.
   1. Group which will receive L. reuteri at a dose 100.000.000 CFU per dose plus lactulose in a dose 1-3 ml/kg, according to the stool frequency and consistency, for 3 months.
   2. Group which will receive placebo plus lactulose in a dose 1-3 ml/kg, according to the stool frequency and consistency, for 3 months.

   All children with a presence of a impacted stool in rectum (on digital rectal exam) at baseline will receive bisacodyl suppository for disimpaction. As a part of randomized, double blind controlled trail, patients will be randomized into one group (A or B) and none of investigators or patients will know true nature of the product (active product or placebo).
4. Hypothesis L. reuteri may effectively treat chronic constipation in children.
5. Aims To evaluate the effect of L. reuteri on the frequency and consistency of stools and episodes of pain in children with chronic constipation
6. Randomization: as in Part I.

BASELINE (VISIT 1): randomization According to the list of patients they will be randomized into two groups (A or B): "probiotic" group and "placebo" group.

VISIT 2: 4 weeks after randomization. END OF STUDY (VISIT 3): End of study 3 months after baseline. VISIT 4: 4 weeks after the end of study (16 weeks after the baseline).

All the symptoms will be monitored using diaries attached to protocol.

ETHICS: as in Part I.

ADHERENCE: as in Part I.

ELIGIBILITY:
Inclusion Criteria:

* Children with functional abdominal pain (age 4-18 years)
* Children with chronic constipation (age 2-18 years)

Exclusion Criteria:

* Immunodeficiency
* Receiving probiotic and/or prebiotic products 7 days prior to enrolment
* Neoplasms
* Chronic disorders
* Presence of "red flags":

  * Weight loss of more than 10%
  * Growth retardation or growth failure
  * Extraintestinal symptoms (fever, rash, joint pain, aphthae, affection of the urinary system)
  * Frequent vomiting
  * Abnormalities in laboratory findings (anemia, elevated ESR)
  * Abnormalities in clinical findings (organomegaly, perianal disease)

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-06 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Intensity of abdominal pain | 3 months
  Pain score on visual-analogue scale during treatment
Severity of chronic constipation | 3 months
  Stool consistency score on Bristol stool scale during treatment

SECONDARY OUTCOMES:
Intensity of abdominal pain after treatment | 1 month
  Pain score on visual-analogue scale in a period of 1 month after stopping treatment
Severity of chronic constipation after treatment | 1 month
  Stool consistency score on Bristol stool scale in a period of 1 month after stopping treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sanja Kolaček, MD, PhD, Principal Investigator — Head, Department of Pediatrics, Clinical Professor; Iva Hojsak, MD, PhD, Study Director — Consultant in Pediatric Gastroenterology; Oleg Jadrešin, MD, MSc, Study Chair — Consultant in Pediatric Gastroenterology
Locations (1):
- University Hospital Centre "Sisters of Mercy", Zagreb, Croatia

REFERENCES:
- [Background] Savino F, Cordisco L, Tarasco V, Palumeri E, Calabrese R, Oggero R, Roos S, Matteuzzi D. Lactobacillus reuteri DSM 17938 in infantile colic: a randomized, double-blind, placebo-controlled trial. Pediatrics. 2010 Sep;126(3):e526-33. doi: 10.1542/peds.2010-0433. Epub 2010 Aug 16. PMID 20713478
- [Background] Coccorullo P, Strisciuglio C, Martinelli M, Miele E, Greco L, Staiano A. Lactobacillus reuteri (DSM 17938) in infants with functional chronic constipation: a double-blind, randomized, placebo-controlled study. J Pediatr. 2010 Oct;157(4):598-602. doi: 10.1016/j.jpeds.2010.04.066. Epub 2010 Jun 12. PMID 20542295
- [Background] Szajewska H. Probiotics and functional gastrointestinal disorders. J Pediatr Gastroenterol Nutr. 2011 Dec;53 Suppl 2:S30-2. No abstract available. PMID 22235462
- [Background] Tabbers MM, Chmielewska A, Roseboom MG, Crastes N, Perrin C, Reitsma JB, Norbruis O, Szajewska H, Benninga MA. Fermented milk containing Bifidobacterium lactis DN-173 010 in childhood constipation: a randomized, double-blind, controlled trial. Pediatrics. 2011 Jun;127(6):e1392-9. doi: 10.1542/peds.2010-2590. Epub 2011 May 23. PMID 21606153
- [Background] Horvath A, Dziechciarz P, Szajewska H. Meta-analysis: Lactobacillus rhamnosus GG for abdominal pain-related functional gastrointestinal disorders in childhood. Aliment Pharmacol Ther. 2011 Jun;33(12):1302-10. doi: 10.1111/j.1365-2036.2011.04665.x. Epub 2011 Apr 20. PMID 21507030
- [Background] Chmielewska A, Szajewska H. Systematic review of randomised controlled trials: probiotics for functional constipation. World J Gastroenterol. 2010 Jan 7;16(1):69-75. doi: 10.3748/wjg.v16.i1.69. PMID 20039451
- [Background] Gawronska A, Dziechciarz P, Horvath A, Szajewska H. A randomized double-blind placebo-controlled trial of Lactobacillus GG for abdominal pain disorders in children. Aliment Pharmacol Ther. 2007 Jan 15;25(2):177-84. doi: 10.1111/j.1365-2036.2006.03175.x. PMID 17229242
- [Background] Szajewska H, Setty M, Mrukowicz J, Guandalini S. Probiotics in gastrointestinal diseases in children: hard and not-so-hard evidence of efficacy. J Pediatr Gastroenterol Nutr. 2006 May;42(5):454-75. doi: 10.1097/01.mpg.0000221913.88511.72. PMID 16707966
- [Derived] Jadresin O, Sila S, Trivic I, Misak Z, Hojsak I, Kolacek S. Lack of Benefit of Lactobacillus reuteri DSM 17938 as an Addition to the Treatment of Functional Constipation. J Pediatr Gastroenterol Nutr. 2018 Dec;67(6):763-766. doi: 10.1097/MPG.0000000000002134. PMID 30134331
- [Derived] Jadresin O, Hojsak I, Misak Z, Kekez AJ, Trbojevic T, Ivkovic L, Kolacek S. Lactobacillus reuteri DSM 17938 in the Treatment of Functional Abdominal Pain in Children: RCT Study. J Pediatr Gastroenterol Nutr. 2017 Jun;64(6):925-929. doi: 10.1097/MPG.0000000000001478. PMID 27906800